CLINICAL TRIAL: NCT01872832
Title: A Phase 1, Randomized, Single-Blind, Placebo-Controlled Study to Evaluate Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of Single and Multiple Doses of RDEA3170 in Healthy Male Japanese Subjects
Brief Title: Single and Multiple Dose Study in Japanese Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Ardea Biosciences, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: RDEA3170-104
Record Dates: First submitted 2013-06-03; First posted 2013-06-07 (Estimated); Last update posted 2014-01-09 (Estimated); Status verified 2014-01

CONDITIONS: Gout
MeSH Terms: conditions — Gout | interventions — verinurad

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (4):
- 5 mg RDEA3170 (Experimental): RDEA3170 5 mg or placebo fasted and fed
  Interventions: Drug: RDEA3170 and Placebo
- 10 mg RDEA3170 (Experimental): RDEA3170 10 mg or placebo fasted and fed
  Interventions: Drug: RDEA3170 and Placebo
- 15 mg RDEA3170 (Experimental): RDEA3170 15 mg or placebo fasted and fed
  Interventions: Drug: RDEA3170 and Placebo
- 2.5 mg RDEA3170 (Experimental): RDEA3170 2.5 mg or placebo fasted and fed
  Interventions: Drug: RDEA3170 and Placebo

INTERVENTIONS:
Drug: RDEA3170 and Placebo

SUMMARY:
This study will explore the safety, tolerability, and serum uric acid lowering effect of RDEA3170 in healthy Japanese males to allow comparison with the Western population.

DETAILED DESCRIPTION:
While clinical studies of RDEA3170 to date have been limited to a Western population, it is recognized that both intrinsic and extrinsic factors may impact the PK, PD, safety, and dose response in different ethnic populations. The purpose of this study is to explore the safety, tolerability, pharmacokinetic (PK), and pharmacodynamic (PD) of single and multiple doses of RDEA3170 in healthy Japanese males, and to allow comparison of these parameters with the Western population.

ELIGIBILITY:
Inclusion Criteria:

* Able to understand the study procedures and the risks involved, and willing to provide written informed consent before the first study related activity.
* Healthy adult male subject born in Japan.
* Subject has parents and grandparents who are Japanese.
* Subject is in possession of a valid Japanese passport.
* All laboratory parameters should be within normal limits or considered not clinically significant by the investigator.
* Screening serum urate level ≥ 4.5 mg/dL.
* Subject is free of any clinically significant disease that requires a physician's care and/or would interfere with study evaluations or procedures.
* Subject has a normal or clinically acceptable physical examination.
* Subject has no clinically relevant abnormalities in blood pressure, heart rate, and body temperature, per the Investigator's judgment.

Exclusion Criteria:

* Positive serology to human immunodeficiency virus (HIV-1 or HIV-2).
* Positive test for active hepatitis B or hepatitis C infection.
* History or suspicion of kidney stones.
* Undergone major surgery within 3 months prior to Day 1.
* Exposed to an investigational drug (or a medical device) within 30 days or 5 half-lives of the investigational drug (whichever is longer) prior to Day 1 or is currently participating in another study of an investigational drug (or medical device).
* Prior exposure to RDEA3170.

Ages: 20 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 46 (Actual)
Dates: Start 2013-06; Primary Completion 2013-09 (Actual); Study Completion 2013-11 (Actual)

PRIMARY OUTCOMES:
Incidence of Adverse Events and Changes in Laboratory, Electrocardiogram, and Vital Signs Parameters | 5 to 6 weeks
PK profile of RDEA3170 from plasma and urine | Day 1 through 15
  Profile in terms of AUC, Tmax, Cmax, and t1/2
  AUC: area under the plasma concentration versus time curve; Tmax: time to maximum plasma concentration; Cmax: maximum plasma drug concentration; t1/2: apparent terminal half-life
PD profile of RDEA3170 from serum and urine | Day 1 through 15
  Profile in terms of sUA concentration; CLr; urine uric acid excretion amount; fractional excretion of uric acid
  sUA: serume urate; CLr: renal clearance

CONTACTS AND LOCATIONS:
Overall Officials: S Baumgartner, MD, Study Director — Ardea Biosciences, Inc.
Locations (1):
- Glendale, California, United States